CLINICAL TRIAL: NCT06995872
Title: Phase I Trial of rhIL-15 Plus Dinutuximab Plus Irinotecan/Temozolomide for Children and Young Adults With Relapsed/Refractory Neuroblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001842; 001842-C
Record Dates: First submitted 2025-05-28; First posted 2025-05-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08-18

CONDITIONS: Neuroblastoma
Keywords: Irinotecan; Temozolomide; ch14.18; IL-15; Neuroblastoma; Dinituximab
MeSH Terms: conditions — Neuroblastoma | interventions — Temozolomide; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Participants will receive dinutuximab at a dose of 17.5 mg/m2/day x 4 days, in combination with escalating doses of rhIL-15 and fixed dose irinotecan and temozolomide.
  Interventions: Drug: rhIL-15; Drug: Dinituximab; Drug: Temozolomide; Drug: Irinotecan Hydrochloride

INTERVENTIONS:
Drug: rhIL-15 — rhIL-15 will be given at a dose of 0.13-2 mcg/kg/day (based on dose level) as a continuous IV infusion for 5 days each cycle.
Drug: Dinituximab — Dinituximab will be given at a dose of 17.5 mg/m^2/dose by IV on days 2-5 of each cycle.
Drug: Temozolomide — Temozolomide will be given orally (PO) at a dose based on weight on days 1-5 of each cycle beginning with cycle 2.
Drug: Irinotecan Hydrochloride — Irinotecan will be given at a dose of 50 mg/m^2/dose by IV on days 1-5 of each cycle beginning with cycle 2.

SUMMARY:
Background:

Neuroblastoma is a type of cancer that causes tumors in nerves. It affects mainly infants and toddlers, and it causes about 15 percent of cancer-related deaths in children.

Objective:

To test a new drug (rhIL-15), combined with 3 standard cancer drugs, in people with neuroblastoma.

Eligibility:

People aged 3 to 35 years with neuroblastoma that did not respond or returned after standard treatment.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests. They will have imaging scans and tests of their heart and lungs. They will have a bone marrow biopsy: A sample of tissue and fluid from inside a bone will be removed with a large needle.

Participants will be treated in 21-day cycles. They may have up to 4 treatment cycles.

rhIL-15 is given through a needle into a vein over 5 to 7 days during the first week of each cycle. Participants will stay in the hospital while they are receiving the rhIL-15.

Starting in the second week of the second cycle, participants will receive other drugs for treating cancer. They will have no study treatments during the third week of each cycle.

Participants will visit the clinic at least 2 times a week throughout all 4 treatment cycles. They will have a physical exam and blood tests during these visits. Imaging scans, bone marrow biopsy, and other tests will be repeated at the end of cycles 2 and 4.

Participants will have a follow-up visit 6 months after treatment ends. This visit will include a physical exam with blood and urine tests.

DETAILED DESCRIPTION:
BACKGROUND:

Neuroblastoma is the most common extracranial pediatric solid tumor, accounting for approximately 15 percent of all childhood cancer-related deaths. Neuroblastoma predominantly affects infants and toddlers and manifests as a solid tumor of the parasympathetic ganglia. Despite multi-modal therapy including multiagent induction chemotherapy, surgery, consolidation with tandem autologous bone marrow transplantation, radiation, anti-GD2 antibody therapy plus GMCSF, and differentiation therapy with cis-retinoic acid, less than 30 percent of newly-diagnosed patients with high-risk neuroblastoma attain long-term remissions, highlighting the need for new and more effective therapies. Based on our preclinical studies, we are proposing in this study, to evaluate recombinant human interleukin (IL)-15 (rhIL-15) with the FDA-approved anti-GD2 antibody, dinutuximab, and chemotherapy (i.e., irinotecan and temozolomide) in children with relapsed/refractory neuroblastoma with the goal to evaluate the safety, toxicity and RP2D of rhIL-15 as part of this chemo-immunotherapy regimen.

OBJECTIVES:

* Primary Objective

  -- Assess the safety of rhIL-15 combined with dinutuximab and irinotecan/temozolomide in pediatric and young adult participants with recurrent or refractory neuroblastoma by determining the recommended phase 2 dose (RP2D) based on dose-limiting toxicity (DLT) of defined adverse events (AEs).
* Secondary Objectives

  * Assess the preliminary anti-tumor activity of rhIL-15 when added to a regimen with dinutuximab/temozolomide/irinotecan in children and young adults with relapsed and/or refractory neuroblastoma.
  * Assess the pharmacokinetics of rhIL-15 when given with dinutuximab.
* Exploratory Objectives

  * Determine the function and kinetics of natural killer (NK) cells and CD8 T cells in the peripheral blood after therapy with rhIL-15 and dinutuximab.
  * Determine if plasma cell free DNA (cfDNA) correlates with tumor burden and response
  * Evaluate tumor heterogeneity pre/post chemo-immunotherapy in bone marrow samples if tumor present.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Disease Requirements:

  * Histologic diagnosis: Participants must have pathology-confirmed neuroblastoma (no time limit). Old reports and tissue blocks can be used if available. Confirmation of disease will be based on the review of pathology at the NIH any time before starting and is based on one of the following: (1) A confirmed pathological diagnosis made from tumor tissue by light microscopy (with or without immunohistology or electron microscopy), (2) the combination of bilateral bone marrow aspirate and trephine biopsy containing confirmed tumor cells (e.g., syncytia or immunocytologically positive clumps of cells) and increased levels of urinary catecholamine metabolites.
  * Active disease status: Participants must have relapsed and/or refractory disease after receiving frontline chemotherapy and at least one salvage treatment (can include dinutuximab, temozolomide, and/or irinotecan), with no alternative curative options.
  * Documentation of disease: Participants must have evaluable disease according to the International Neuroblastoma Response Criteria (INRC). This means they must have an area of active disease that can be identified by MIBG, PET, MRI/CT, or bone marrow studies. Participants must have at least ONE of the following at the time of enrollment:

    * Measurable tumors on magnetic resonance imaging (MRI) or computed tomography (CT) scan. Measurable is defined as >=10 mm in at least one dimension.
    * 123MIBG-avid lesion detected on 123MIBG scan with positive uptake at a minimum of one site. This site must represent disease recurrence after completion of therapy, progressive disease on therapy, or refractory disease during induction.
    * Participants with resistant/refractory soft tissue disease that is not 123MIBG avid or does not demonstrate increased FDG uptake on PET scan must undergo a biopsy to document the presence of viable neuroblastoma. Biopsy is not required for participants who have a new site of soft tissue disease (radiographic evidence of disease progression) regardless of whether progression occurs while receiving therapy or after completion of therapy.
    * Participants with bone marrow disease in at least one sample from bilateral bone marrow biopsies will be eligible (documented neuroblastoma cells).
    * Participants with a history of CNS disease must have no clinical or radiological evidence of active CNS disease at the time of study enrollment.
* Prior Therapy:

Potential trial participants should have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment.

* Chemo-immunotherapy: Participants are eligible if they have received prior therapy with dinutuximab/temozolomide/irinotecan, even if they may not have responded previously
* Myelosuppressive chemotherapy: Potential trial participants should have recovered from clinically significant myelosuppression.
* Non-chemotherapy anti-neoplastic agents: With anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or ANC counts), sufficient time needs to have passed for the drug to have cleared the body. This is to prevent overlapping non-hematological toxicity.
* Anti-GD2 antibody: toxicity related to prior antibody therapy must be recovered to grade <=1.
* Radiation therapy: Given the possible negative effect of radiation on bone marrow cells and count recovery after chemotherapy, potential trial participants should have recovered from clinically significant radiation-induced myelosuppression. Palliative radiation while on study is not permitted.
* Stem cell transplants (SCT): After autologous stem cell transplants or stem cell infusions (including stem cell infusions given as supportive care following 131 I-MIBG therapy), all hematologic and other eligibility criteria must have been met.
* 131I-MIBG therapy: After therapeutic 131 I-MIBG, all hematologic and other eligibility criteria must have been met.
* Participants who have received drugs that are strong inducers or inhibitors of CYP3A4 within 7 days before study enrollment are not eligible.

  -Age Requirement:
* Age >= 3 years and <= 35 years at the time of enrollment.

  -Clinical Performance Status:
* Participants >= 16 years of age: Karnofsky >= 50 percent; Participants < 16 years of age: Lansky scale >= 50 percent. Participants who are unable to walk because of paralysis, but who are upright in a wheelchair will be considered ambulatory to calculate the performance score.

  -Adequate Organ and Marrow Function as Defined Below:
* Absolute neutrophil count: >= 1000/mcL
* Platelets: >= 100,000/mcL (transfusion-independent)
* Total bilirubin: <=2 X ULN (except in the case of participants with documented Gilbert s disease < 3x ULN)
* AST(SGOT)/ALT(SGPT): <=3 X institutional upper limit of normal
* Creatinine: <= the maximum for age listed in the table below OR
* Measured creatinine clearance: >= 60 mL/min/1.73 m^2 for participants with creatinine levels above the max listed below per age:

  * Age (Years) <=5, Maximum Serum Creatinine <= 0.8 (mg/dL)
  * Age (Years) 6 to <= 10, Maximum Serum Creatinine <=1.0 (mg/dL)
  * Age (Years) >10, Maximum Serum Creatinine <= 1.2 (mg/dL)
* Cardiac function: Left ventricular ejection fraction >= 52 percent.
* Pulmonary Function

  * Baseline oxygen saturation >92 percent on room air at rest
  * Participants with respiratory symptoms clinically concerning for decreased pulmonary function must have a DLCO/adjusted > 45 percent. For children who are unable to cooperate for PFTs, they must not have dyspnea at rest or a known requirement for supplemental oxygen.

    * Given the teratogenic effects of the therapy, participants of childbearing or child fathering potential must agree to be abstinent or use highly effective contraception (hormonal; intrauterine device; surgical sterilization). This restriction will be from the time of enrollment on this study and for four months (in persons who can father children) or six months (in participants who can bear children) after completing therapy. Participants may also confirm with their partners that they are using a highly effective method.
    * Participants who are nursing or plan to nurse must agree to discontinue/postpone nursing while on study therapy since it cannot be ruled out with certainty that any of the investigational drugs can be transmitted via breast milk.
    * Ability of participant or parents/legal guardian to understand and sign a written informed consent document.

EXCLUSION CRITERIA:

* Presence of pericardial effusion.
* Current/active human immunodeficiency virus (HIV) infection, as measured by seropositivity for HIV antibody.
* Current/active HBV/HCV infection as measured by seropositivity for Hepatitis C or positive for Hepatitis B surface antigen (HBsAg).
* History of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biological composition to irinotecan and temozolomide used in study.
* Participants with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous.
* Positive serum or urine beta-HCG pregnancy test performed at screening due to the teratogenic effects of chemotherapy.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants must not have >= grade 2 diarrhea at the time of entry.
* Participants who are unable to tolerate oral/nasogastric/gastrostomy medications will not be eligible for this trial. Additionally, participants with significant malabsorption will not be eligible for this trial.
* Participants must not have uncontrolled infection.
* Participants with a history of Grade 4 allergic reactions to anti-GD2 antibodies or reactions that required permanent discontinuation of the anti-GD2 therapy are not eligible.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and determine the MTD of rhIL-15 combined with dinutuximab/temozolomide/irinotecan | 6 weeks
  Assessment of AEs and DLTs in participants.

SECONDARY OUTCOMES:
Anti-tumor activity | 6 months
  Response will be evaluated by applying the INRC after even numbers of cycles. This includes response at the following sites: Primary tumor, metastatic soft tissue and bone site, bone marrow.
Pharmacokinetics | 3 weeks
  rhIL-15 levels in the plasma of participants at various timepoints after initiation of the rhIL-15 infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ha Rosa Nguyen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC.
Access Criteria: The scientific data will be findable by key words or MeSH terms used during publication of manuscripts.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001842-C.html